CLINICAL TRIAL: NCT07315139
Title: Effect of Pentoxifylline on Inflammatory Markers in Non-Diabetic Chronic Kidney Disease Patients
Brief Title: Pentoxifylline on Inflammatory Markers in Non-Diabetic Chronic Kidney Disease Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ashraf Hassan, Assistant Professor of Internal Medicine and Nephrology, Faculty of Medicine, Ain shams University, Cairo, Egypt., Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMASU MS 53/2023
Record Dates: First submitted 2025-12-18; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Pentoxifylline; Inflammatory Markers; Non-Diabetic; Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Angiotensin-Converting Enzyme Inhibitors; Ramipril; Pentoxifylline

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): Patients received the standard therapy. The routine standard consisted of angiotensin-converting enzyme inhibitors (ACEI) (Ramipril 1.25 mg), a calcium-based phosphate binder (calcium acetate 700 mg, containing 180 mg of calcium), alfacalcidol (0.25 µg), antihypertensive medications, and diuretics.
  Interventions: Drug: Angiotensin-converting enzyme inhibitors (Ramipril)
- Group 2 (Experimental): Patients received one capsule of Pentoxifylline 400 mg twice daily for 6 months, in addition to their standard therapy.
  Interventions: Drug: Pentoxifylline

INTERVENTIONS:
Drug: Angiotensin-converting enzyme inhibitors (Ramipril) — Patients received the standard therapy. The routine standard consisted of angiotensin-converting enzyme inhibitors (ACEI) (Ramipril 1.25 mg), a calcium-based phosphate binder (calcium acetate 700 mg, containing 180 mg of calcium), alfacalcidol (0.25 µg), antihypertensive medications, and diuretics.
  Arms: Group 1
Drug: Pentoxifylline — Patients received one capsule of Pentoxifylline 400 mg twice daily for 6 months, in addition to their standard therapy.
  Arms: Group 2

SUMMARY:
This study aimed to determine the impact of Pentoxifylline on inflammatory biomarkers and the progression of chronic kidney disease in non-diabetic patients.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) is a progressive condition that affects >10% of the general population worldwide, amounting to >800 million individuals.

The diagnosis of CKD is established by laboratory testing, most often by estimating glomerular filtration rate (GFR) from a filtration marker, such as serum creatinine or cystatin C, using various formulas, or by testing urine for albumin or protein (or both).

Pentoxifylline (PTX), a synthetic dimethylxanthine derivative used initially to treat intermittent claudication in patients with peripheral arterial disease due to its hemorheological effects, has been shown to have potent antioxidant, anti-inflammatory, antidiabetic, anti-cellular-damage, and antifibrotic effects.

ELIGIBILITY:
Inclusion Criteria:

* Age ˃ 18 years old.
* Both sexes.
* Patients with chronic kidney disease (CKD) stages G3, G4.
* Patients with proteinuria < 1 g.

Exclusion Criteria:

* Patients who are terminally ill.
* Patients with Diabetes mellitus.
* Patients with proteinuria > 1 g.
* Patients with a history of hemodialysis.
* Patients with active infection or hospitalized.
* Patients with recent cerebral and /or retinal Hemorrhage.
* Patients taking warfarin or theophylline-containing drugs.
* women who are taking oral contraceptives, pregnant, or lactating
* Patients with a history of adverse reactions to Pentoxifylline.
* Patients with polycystic kidney disease.
* Patients with obstructive uropathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Levels of inflammatory marker | 3 months post-procedure
  Levels of inflammatory marker was recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.